CLINICAL TRIAL: NCT07033156
Title: An Exploratory Study on Gene Methylation Detection of Colorectal Cancer（CRC）
Brief Title: An Exploratory Study on Gene Methylation Detection of Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Jinjiang Central Hospital (Unknown); Xilingol League Central Hospital (Unknown); Zybio Inc. (Unknown); Haining Central Hospital (Unknown); Tiantai County People's Hospital (Unknown); Xianju County People's Hospital (Unknown); Fuyang District People's Hospital (Unknown); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhenyuan Qian, associate senior doctor, Zhejiang Provincial People's Hospital
Other Study IDs: QT2024274
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: CRC (Colorectal Cancer); Adenoma Colon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: This study does not require intervention trials — This study does not require intervention trials

SUMMARY:
The goal of this exploration study is to evaluate the performance of a colorectal cancer (CRC) early screening model based on the DNA methylation technology platform. The study focuses on individuals over the age of 40 and aims to identify and verify methylation biomarkers for colorectal cancer using stool samples . The main question it aims to answer is:

Can a DNA methylation-based model effectively detect colorectal cancer and adenoma in individuals over 40 using non-invasive stool samples?

Participants will provide stool samples for methylation analysis. The study results will be used solely for internal product performance evaluation and optimization by the sponsor and will not be used for product registration or influence any clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Sample Source: Hospital physical examination, outpatient, and inpatient patients;
2. Patient Information: Patient information (such as age, hospital ID number, gender, clinical diagnosis, colonoscopy and pathology results) is traceable;
3. Age Requirement: ≥ 40 years old;
4. Sampling Time Requirement: Stool and plasma samples must be collected within 3 months prior to colonoscopy (stool samples are preferred).

Exclusion Criteria:

1. Unclear Sample Collection Information: Samples with unclear collection time, or stool samples not collected within 3 months prior to colonoscopy, or samples with incomplete clinical information that cannot be traced;
2. Non-compliance with Sample Requirements: Samples that do not meet the collection and storage requirements;
3. History of Disease: Subjects with a history or treatment of colorectal cancer (CRC) or advanced precancerous lesions;
4. Insufficient Sample Volume: Samples with insufficient volume that cannot meet the requirements of the assessment system testing;
5. Hereditary Diseases: Subjects with a diagnosis or family history of the following diseases:Familial adenomatous polyposis (FAP), including attenuated FAP and Gardner syndrome;Hereditary nonpolyposis colorectal cancer syndrome (HNPCC or Lynch syndrome);Other hereditary cancer syndromes, including but not limited to Peutz-Jeghers syndrome, MYH-associated polyposis (MAP), Turcot syndrome (or Crail syndrome), Cowden syndrome, juvenile polyposis, neurofibromatosis, or familial proliferative polyposis (FAP);
6. Inflammatory Bowel Disease (IBD): Subjects with a diagnosis or personal history of IBD, including chronic ulcerative colitis and/or Crohn's disease;
7. Cronkhite-Canada Syndrome: Subjects with a diagnosis of Cronkhite-Canada syndrome.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital physical examination, outpatient, and inpatient patients;
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
human stool gene methylation | 2024.12-2025.8
  The core of the study is to detect the methylation levels of three genes in human stool samples. These three genes are SDC2, COL4A2, and C9orf50. The procedure includes stool sample collection, stool nucleic acid extraction, bisulfite conversion, and detection using the qMSP (quantitative Methylation-Specific PCR) method.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No